CLINICAL TRIAL: NCT04380896
Title: COVID-19 Staff Testing of Antibody Responses Study (CO-STARS)
Acronym: Co-Stars
Status: Completed | Type: Observational
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20CB17
Record Dates: First submitted 2020-05-04; First posted 2020-05-08 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Each sample will be tested using the EDITM diagnostic assay which detects the optical density of antibodies in serum samples to the nucleo-capsid protein SARS-CoV-2. Both IgM and IgG antibodies to the nucleo-capsid protein will be tested and reported.
  At the end of the study the samples will be stored at -70oC in the freezers of the Great Ormond Street Camelia Botnar Laboratories for future research. Future studies may involve genetic testing on the samples and this has been highlighted on the consent form.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SARS-CoV-2 Seropositive Cases: It will be formed of approximately N= 200 to 350 staff members
  Core Group of PCR Confirmed Cases N ~ 150 to 250:
  A) Symptoms consistent with SARS-CoV-2 infection and SARS-CoV-2 PCR Positive N ~ 150 to 250 OR
  Other SARS-CoV-2 Sero-positives N ~ 50 to 100:
  B) Symptoms consistent with SARS-CoV-2 infection and SARS-CoV-2 PCR Negative cases. OR C) No symptoms consistent with SARS-CoV-2 infection and PCR Not Tested cases
  Interventions: Other: Blood test; Other: Standardised questionnaires
- SARS-CoV-2 Seronegative Comparison Group: It will be formed of approximately N= 800 to 900 staff members
  Core Comparison Group N ~ 800 A) Have not had clinical symptoms consistent with SARS-CoV-2 infection OR
  Other Seronegatives N ~ 100 B) Have had sympoms of SARS-CoV-2 infection but have been tested and were PCR positive or negative but have not developed antibodies at 21 days
  Interventions: Other: Blood test; Other: Standardised questionnaires

INTERVENTIONS:
Other: Blood test — Blood tests (8ml in total) 4ml blood for serological testing (measure the antibody titres to the SARS-CoV-2 nucleo-capsid protein (4ml) and 4ml EDTA to be stored for future research will be taken for each group.
Other: Standardised questionnaires — It will be an online questionnaire about staff members health, symptoms of SARS-CoV-2 and contact with SARS-CoV-2. All participants will also be asked to complete a detailed symptom and electronic questionnaire prior to each appointment.

SUMMARY:
This study will perform prospective repeated serological antibody testing on a cohort of at least 1000 healthcare workers at Great Ormond Street Hospital. Within this cohort, a subset of 150-250 staff members with confirmed (PCR positive) SARS-CoV-2 disease will be followed with intensive monthly testing for 6 months to determine whether antibody levels in the blood are maintained or decrease during this time. All 1000 recruited healthcare workers will be followed 6-monthly

DETAILED DESCRIPTION:
A total of 250 healthcare workers are currently off sick with symptoms of SARS-CoV-2 infection (COVID-19) while 99 additional members of staff have been diagnosed with confirmed SARS-CoV-2 at Great Ormond Street Hospital. As a consequence, all routine surgery, out-patient activity and day cases have been postponed or cancelled altogether. It is therefore critical for us to understand whether or not this disease will continue to threaten staff health or whether natural infection will give rise to long lasting immunity.

This is a 2-arm prospective cohort study recruiting at least 1000 healthcare workers at GOSH over 6 years.Staff will be recruited and coordinated from each department to be representative of the full diversity of healthcare workers at the Trust. The age distribution of the participants will be monitored on a weekly, basis against the known age distribution of the hospital to ensure that the sample is representative.

Trust communications team will send an all staff email to inform them about this research project asking them to get in touch with the study team if they wish to participate and they meet the basic eligibility criteria. Potential participants will be asked voluntarily to attend a face to face appointment in person (or if preferred by telephone or 1:1 video teleconference meeting) to enable trained study staff to seek informed consent before they enter the study. Informed consent will be undertaken by study staff who are Good Clinical Practice trained, Human Tissue Act trained, study trained, GOSH consent trained and registered in the study log.

The consent process will specifically cover the reason for the study, the storage of samples and agreement for future samples to be tested once improved testing is made available. Once the member of staff has provided informed consent, they will be asked to undertake an online questionnaire in which they will record demographic details including age, sex, email address and telephone contact for results and coordinating follow up. The questionnaire will also record details of SARS-CoV-2 like symptoms, contact with SARS-CoV-2, pre-existing co-morbidities and medication or treatments that may interfere with serological testing.

After providing informed consent, the staff members then be asked attend the study phlebotomy testing clinic. Appointments will be 20 minutes in length but actual blood sampling for serological testing will be 5-10 minutes to allow plenty of time and space for staff members to be tested to maintain social distancing. A total of 8ml of blood will be stored for testing.

Follow up sampling and questionnaires of approximately 200 staff members with PCR confirmed SARS-CoV-2 infected staff will take place monthly. While follow up of all ~800 asymptomatic staff members will take place 6 monthly. All staff will continue to have access to the GOSH PCR COVID19 testing program (as they do at present). This will enable us to confirm with PCR testing any new (or reinfected) positive staff member with COVID-19 over the duration of the study.

When initially asymptomatic seronegative staff become serologically positive during the course of the study, they will remain under active surveillance but they will switch arms of the study and they will contribute to the active follow up of serologically positive patients.

If staff leave the GOSH NHS trust during the study they will still be eligible to remain in the study and be followed up and we will update their contact details on the follow-up questionnaire.

After the initial intensive phase, all approximately 1000 recruits will be followed 6 monthly for the 6 year duration of the study. Follow-up visits will be arranged following the baseline assessment. The same blood tests 4ml EDTA and 4ml serum will be taken at each follow up appointment as well as the same symptom questionnaire.

ELIGIBILITY:
Inclusion Criteria for ARM 1: SARS-CoV-2 Seropositive Cases:

* Healthcare worker at GOSH
* >18 years of age
* ALL have confirmed detectable antibodies to SARS-CoV-2 infection on baseline screen

Then can be recruited into either of the following sub-groups

1. Core Group of PCR Confirmed Cases : Must have symptoms consistent with SARS-CoV-2 infection and SARS-CoV-2 PCR Positive
2. Other SARS-CoV-2 Sero-positives: May have Symptoms consistent with SARS-CoV-2 infection and SARS-CoV-2 PCR Negative cases OR May have no symptoms consistent with SARS-CoV-2 infection and PCR Not Tested cases

Inclusion Criteria for ARM 2: SARS-CoV-2 Seronegative Comparison Group :

* Healthcare worker at GOSH
* >18 years of age
* ALL have confirmed negative antibodies to SARS-CoV-2 infection on baseline screen

Then can be recruited into either of the following Sub-groups:

1. Core Comparison Group: Have not had clinical symptoms consistent with SARS-CoV-2 infection*
2. Other Seronegatives: Have had symptoms of SARS-CoV-2 infection but have been tested and were PCR positive or negative but have not developed antibodies at 21 days

   * Clinical Symptoms for SARS-CoV-2 infection are defined as one of:

1) New and persistent cough 2) Confirmed temperatures of 37.8 and above 3) Anosmia

General Exclusion Criteria :

* <18 years of age
* On immunosuppressive or immunomodulatory medication that may impact test reliability
* Received any blood product including immunoglobulins after October 2019
* Has received convalescent sera as treatment
* Current diagnosis of a malignancy that may impact test reliability
* Those lacking capacity to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population will comprise frontline healthcare workers selected to be representative of all departments at Great Ormond Street Hospital. The researcher will ensure that equal numbers of men and women are recruited from each department and that age ranges are representative of the trust population age distribution.We will also check the age distribution of the participants on a weekly basis during recruitment against the known age distribution of the hospital to ensure that our sample is representative. If significant differences among ages between the study population and the hospital population age range emerge then we will actively recruit from those age ranges that we have inadequately sampled.
Sampling Method: Probability Sample
Enrollment: 3502 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
Change in serial monthly log-transformed antibody titre levels as measured | 6 months period post infection
  To determine the kinetics (rate of change) of SARS-CoV-2 nucleo-capsid protein antibody titres in proven cases of SARS-CoV-2 over the 6 month period following infection

SECONDARY OUTCOMES:
Proportion of completely asymptomatic healthcare workers with evidence of SARS-CoV-2 antibodies | 12 months
  To determine the proportion of completely asymptomatic healthcare workers who have evidence of SARS-CoV-2 antibodies in their serum indicative of past infection
The attack rate of SARS-CoV-2 in healthcare workers who have antibodies compared to those who do not | Betwen 3 to 6 years
  To determine the attack rate of SARS-CoV-2 in healthcare workers who have antibodies versus those who do not have antibodies
The immune correlates of protection against future exposure to SARS-CoV-2 | Between 3 to 6 years
  To determine the immune correlates of protection (Antibody Titres sufficient for protection) against future exposure to SARS-CoV-2

CONTACTS AND LOCATIONS:
Overall Officials: Louis Grandjean, Dr, Principal Investigator — Great Ormond Street Hospital NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom

REFERENCES:
- [Derived] Lam T, Saso A, Torres Ortiz A, Hatcher J, Woodman M, Chandran S, Thistlethwayte R, Best T, Johnson M, Wagstaffe H, Mai A, Buckland M, Gilmour K, Goldblatt D, Grandjean L; COVID-19 Staff Testing of Antibody Responses (Co-STARs) Study Team. Socioeconomic and Demographic Risk Factors for SARS-CoV-2 Seropositivity Among Healthcare Workers in a UK Hospital: A Prospective Cohort Study. Clin Infect Dis. 2024 Mar 20;78(3):594-602. doi: 10.1093/cid/ciad522. PMID 37647517
- [Derived] Torres Ortiz A, Fenn Torrente F, Twigg A, Hatcher J, Saso A, Lam T, Johnson M, Wagstaffe H, Dhillon R, Mai AL, Goldblatt D, Still R, Buckland M, Gilmour K, Grandjean L. The influence of time on the sensitivity of SARS-CoV-2 serological testing. Sci Rep. 2022 Jun 22;12(1):10517. doi: 10.1038/s41598-022-14351-2. PMID 35732870
- [Derived] Ortiz AT, Torrente FF, Twigg A, Hatcher J, Saso A, Lam T, Johnson M, Wagstaffe H, Dhillon R, Mai AL, Goldblatt D, Still R, Buckland M, Gilmour K, Grandjean L. The Influence of Time on the Sensitivity of SARS-CoV-2 Serological Testing. Res Sq [Preprint]. 2022 Feb 17:rs.3.rs-1286644. doi: 10.21203/rs.3.rs-1286644/v1. PMID 35194596
- [Derived] Grandjean L, Saso A, Torres Ortiz A, Lam T, Hatcher J, Thistlethwayte R, Harris M, Best T, Johnson M, Wagstaffe H, Ralph E, Mai A, Colijn C, Breuer J, Buckland M, Gilmour K, Goldblatt D; COVID-19 Staff Testing of Antibody Responses Study (Co-Stars) team. Long-Term Persistence of Spike Protein Antibody and Predictive Modeling of Antibody Dynamics After Infection With Severe Acute Respiratory Syndrome Coronavirus 2. Clin Infect Dis. 2022 Apr 9;74(7):1220-1229. doi: 10.1093/cid/ciab607. PMID 34218284